CLINICAL TRIAL: NCT04023565
Title: Open-Label Non-Comparative Study of the Effects of a Combination Antihypertensive Treatment With Moxonidine + Perindopril in Hypertensive Patients With Metabolic Syndrome
Brief Title: Moxonidine + Perindopril in Hypertensive Patients With Metabolic Syndrome
Acronym: COMPOSER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sergey V. Nedogoda (Other)
Responsible Party: Sponsor-Investigator, Sergey V. Nedogoda, Dr.Med.Sc., Professor, Volgograd State Medical University
Organization: Volgograd State Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOXOD001
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Arterial Hypertension; Metabolic Syndrome
Keywords: perindopril; moxonidine
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — Perindopril; moxonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- perindopril + moxonidine (Experimental): perindopril 10 mg + moxonidine 0.4 or 0.6 mg a day (given as two divided doses).
  Interventions: Drug: perindopril + moxonidine

INTERVENTIONS:
Drug: perindopril + moxonidine — After 14 days of wash-out period perindopril 10 mg + moxonidine 0.4 mg a day will be prescribed.
  If target BP is achieved after 4 weeks, the dosage will remain unchanged (perindopril 10 mg + moxonidine 0.4 mg a day (given as two divided doses).
  If target BP is not achieved after 4 weeks, the dosage will increase up to perindopril 10 mg + moxonidine 0.6 mg a day (given as two divided doses).

SUMMARY:
The aim of study is to assess the angioprotective effects of antihypertensive combination therapy with perindopril 10 mg and moxonidine 0.4-0.6 mg in patients with arterial hypertension, metabolic syndrome, and obesity, who had Pulse Wave Velocity (PWV) > 10 m/s on the previously administered two-component combination antihypertensive therapy.

Open-label non-comparative prospective study for 24 week for each patient.

DETAILED DESCRIPTION:
According to European Society of Cardiology (ESC) and the European Society of Hypertension (ESH) Guidelines for the management of arterial hypertension 2018 in case of previous combination at full dose does not allow to achieve the target Blood Pressure (BP), that therapy might be switch to different two-drug combination.

The study will enroll 120 hypertensive (Grade 1, 2 Arterial Hypertension (AH): Systolic Blood Pressure (SBP) 140-179 mm Hg and Diastolic Blood Pressure (DBP) 90-109 mm Hg According to ESC/ESH Guidelines 2018) patients with metabolic syndrome who met the inclusion criteria when treated with Angiotensin Converting Enzyme Inhibition(ACEi) /Angiotensin Receptor Blocker (ARB) + hydrochlorothiazide (HCTZ)/indapamide or +amlodipine (30 patients in each group):

1. ACEi (except perindopril) + diuretic (HCTZ or indapamide)
2. ACEi (except perindopril) + amlodipine
3. ARB+ diuretic (HCTZ or indapamide)
4. ARB+ amlodipine

Upon obtaining Inform Consent the previous therapy will be discontinued according to recommendations (gradually or at once).

After 14 days of wash-out period perindopril 10 mg + moxonidine 0.4 mg a day will be prescribed.

If target BP is not achieved after 4 weeks, the dosage will increase up to perindopril 10 mg + moxonidine 0.6 mg a day (given as two divided doses).

FORBIDDEN TREATMENTS:

Any other antihypertensives (calcium antagonists, β-blockers, ACEi except perindopril, ARBs, diuretics) for routine AH management (except those used to resolve the uncontrolled hypertension).

CRITERIA FOR PREMATURE PATIENT WITHDRAWAL FROM THE STUDY:

1. Withdrawal of informed consent by the patient at any time of the study.
2. Need for uncontrolled hypertension management occurring more than 2 times weekly throughout the 2 consecutive weeks during study period.
3. Need for the third antihypertensive drug.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male and female) aging 18 to 70 years.
2. Grade 1, 2 AH (SBP 140-179 mm Hg and/or DBP 90-109 mm Hg according 2018 ESH/ESC guidelines)
3. PWV > 10 m/s
4. Previous two-component antihypertensive therapy (ACEi/ARB+ diuretic (HCTZ or indapamide) or ACEI/ARB + amlodipine) during at least 6 months prior to the study enrollment
5. Metabolic syndrome diagnosed by the 2009 Russian Society of Cardiology (RSC) National Guidelines criteria

   1. THE MAIN SIGN: central (abdominal) obesity defined as waist circumference (WC) above 80 cm in women and above 94 cm in men.
   2. ADDITIONAL CRITERIA:

   i. - arterial hypertension (BP ≥ 130/85 mm Hg) ii. - high triglycerides (≥ 1.7 mmol/l) iii. - decreased HDL-cholesterol (<1.0 mmol/l for men; <1.2 mmol/l for women) iv. - increased LDL-cholesterol > 3.0 mmol/l v. - fasting hyperglycaemia (fasting plasma glucose ≥ 6.1 mmol/l) vi. - impaired glucose tolerance (plasma glucose at 2 hours after glucose load from ≥7.8 to ≤11.1 mmol/l)

   Metabolic syndrome is defined as presence of central obesity and two of the additional criteria.
6. Body Mass Index (BMI) >30 kg/m2.
7. For female patients with childbearing potential: negative pregnancy test and willingness to use reliable methods of contraception until the study treatment completion
8. Voluntarily signed informed consent to participate in the study.

Exclusion Criteria:

1. Contraindications for using ACEi and imidazoline receptor agonists.
2. Administration of perindopril or moxonidine during 6 months before the study onset.
3. Metformin therapy for prophylaxis diabetes mellitus type 2 in patients with pre-diabetes, which had been started within 6 months before the study enrollment. (If a patient receives metformin for a long time, i.e., more than 6 months, he/she can be included in the study, and metformin discontinuation is not required).
4. Statin and/or fibrate therapy started within 6 months before the study enrollment. (If a patient receives statins and/or fibrates for a long time, i.e., more than 6 months, he/she can be included in the study, and discontinuation of statins and fibrates is not required).
5. Current diagnosis of unstable angina, acute and subacute myocardial infarction.
6. Heart failure of any functional class.
7. Grade 3 AH (≥ 180/110 mm Hg).
8. Sinus bradycardia (heart rate ≤50/min).
9. Type 1 or 2 diabetes mellitus.
10. Severe comorbidities, including mental diseases.
11. Acute conditions (infections, exacerbation of chronic diseases, injuries, surgical interventions).
12. Alcohol abuse.
13. Pregnancy and lactation.
14. Serious renal dysfunction (Estimated Glomerular Filtration Rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) ≤30 ml/min/1.73 m2).
15. Serious hepatic dysfunction
16. Malignancies diagnosed and treated during the previous 5 years prior to study enrollment.
17. Inability to understand the study and to give informed consent for participation in it.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pulse wave velocity (PWV) | baseline and 24 weeks
  To assess the PWV after 24 weeks of combination treatment with perindopril 10 mg and moxonidine 0.4-0.6 mg against baseline level.
Change in Central Blood Pressure (BP) | baseline and 24 weeks
  To assess the central BP changes (systolic BP, aortic pulse BP) after 24 weeks of combination treatment with perindopril 10 mg and moxonidine 0.4-0.6 mg against baseline levels.
Change in Reflected wave index | baseline and 24 weeks
  To assess the reflected wave index after 24 weeks of combination treatment with perindopril 10 mg and moxonidine 0.4-0.6 mg against baseline level.

SECONDARY OUTCOMES:
Change in carbohydrate and lipid metabolism parameters markers | baseline and 24 weeks
  To assess the homeostatic model assessment - insulin resistance (HOMA-IR), and lipid metabolism (total cholesterol, triglycerides, low-density lipoprotein (LDL), high-density lipoprotein (HDL)) after 24 weeks of combination treatment with perindopril 10 mg and moxonidine 0.4-0.6 mg against baseline levels.
Change in the adipokine level | baseline and 24 weeks
  To assess the adipokine level (leptin) after 24 weeks of combination treatment with perindopril 10 mg and moxonidine 0.4-0.6 mg against baseline level.
Change in the Inflammatory marker level | baseline and 24 weeks
  To assess the high sensible C-reactive Protein (hs-CRP) after 24 weeks of combination treatment with perindopril 10 mg and moxonidine 0.4-0.6 mg against baseline level.
Change in the renin-angiotensin-aldosterone system hyperactivation marker level | baseline and 24 weeks
  To assess the renin-angiotensin-aldosterone system hyperactivation marker level (plasma aldosterone-to-renin ratio) after 24 weeks of combination treatment with perindopril 10 mg and moxonidine 0.4-0.6 mg against baseline level
Change in the sympathoadrenal system hyperactivation marker levels | baseline and 24 weeks
  To assess the sympathoadrenal system hyperactivation marker levels (urine excretion adrenaline, noradrenaline, dofamine levels) after 24 weeks of combination treatment with perindopril 10 mg and moxonidine 0.4-0.6 mg against baseline levels.
Proportion of patients achieved target BP level | Week 4, Week 12, Week 24
  To assess the proportion of patients (%) achieving target BP levels <130/80 mm Hg at Week 4, Week 12, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V. Nedogoda, Professor, Principal Investigator — Volgograd State Medical University
Locations (1):
- Dept. of Therapy and Endocrinology, Volgograd, Russia